CLINICAL TRIAL: NCT02300779
Title: Randomized Clinical Trial on the Efficacy of an Adapted Bowel Preparation for Diabetic Patients Undergoing a Colonoscopy. DIMEPREP Study
Brief Title: Diet for Colonoscopy Preparation in Diabetic Patients
Acronym: DIMEPREP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Collaborators: Germans Trias i Pujol Hospital (Other)
Responsible Party: Principal Investigator, Marco Antonio Alvarez Gonzalez, MD, Parc de Salut Mar
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: DIMEPREP/PSM/2014
Record Dates: First submitted 2014-11-21; First posted 2014-11-25 (Estimated); Last update posted 2016-04-12 (Estimated); Status verified 2016-04

CONDITIONS: Diabetes Mellitus; Colonic Diseases
Keywords: Colonoscopy; Diabetes Mellitus; Diet; Polyethylene glycols; Efficacy; Personal satisfaction
MeSH Terms: conditions — Diabetes Mellitus; Colonic Diseases; Personal Satisfaction

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low-residue diet (Experimental): Subjects will follow a low-residue diet for 4 days. Their usual treatment for diabetes will be adjusted to the degree of glycemic control.
  Interventions: Dietary Supplement: Low-residue diet
- Usual care (Active Comparator): Subjects will follow a low-residue diet for 3 days (from 4 to 2 days before the procedure) and a liquid diet on the following day (the one before the procedure). No changes in their treatment for diabetes will be made
  Interventions: Dietary Supplement: Usual care

INTERVENTIONS:
Dietary Supplement: Low-residue diet — Subjects will be instructed by members of the research team to follow a low-residue diet for 4 days.
  Bowel cleansing will begin at 9:00 pm on the evening before the colonoscopy is scheduled. Participants will take 8 sachets of the investigational product and take their contents diluted in 2 liters of water. Eight other sachets, also diluted in 2 liters of water will be taken 4 to 5 hours before the procedure.
  Fasting will be required from 2 hours after the bowel cleansing is complete. Their usual treatment for diabetes (whether insulin or an oral agent) will be adjusted.
  Arms: Low-residue diet
Dietary Supplement: Usual care — Subjects will be instructed by members of the research team to follow a low-residue diet for 3 days followed by a liquid-only diet for an additional day.
  Bowel cleansing will begin at 9:00 pm on the evening before the colonoscopy is scheduled. Participants will take 8 sachets of the investigational product and take their contents diluted in 2 liters of water. Eight other sachets, also diluted in 2 liters of water will be taken 4 to 5 hours before the procedure.
  Fasting will be required from 2 hours after the bowel cleansing is complete. No modifications in their usual treatment will be made.
  Arms: Usual care

SUMMARY:
This trial will compare the efficacy of to 2 different sets of dietary recommendations to be followed before colon cleansing for colonoscopy in diabetic patients.

DETAILED DESCRIPTION:
Consecutive diabetic patients undergoing an ambulatory colonoscopy at the participating sites will be randomized to follow one of two different sets of dietary recommendations. The experimental group will be asked to start a low-residue diet 4 days before the procedure, during which the therapy for diabetes will be adjusted. The control group will be asked to follow a low-residue diet for 3 days followed by a liquid diet during the day before the procedure, and no adjustments will be made to their usual treatment.

Colon cleansing will be undertaken with polyethylene glycol (4 liters in the usual split administration scheme) in both groups.

Analogic visual scales and standardized questionnaires on various aspects that may influence the degree of satisfaction about the preparation will be answered by the participants and collected before the colonoscopy. The endoscopist, blinded to the preparation method, will grade the adequacy of the preparation. Adverse events will be recorded up to 1 month after the procedure

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for a diagnostic, screening or follow-up outpatient colonoscopy
* Diabetes mellitus (being treated with insulin or any oral agent).

Exclusion Criteria:

* Unwillingness to participate.
* Hospital admission at the time of colonoscopy.
* Inability to follow instructions
* Active inflammatory bowel disease
* Previous colectomy.
* Incomplete colonoscopies due to technical reasons or contraindication for the procedure as evaluated by the endoscopist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2014-12; Primary Completion 2015-07 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Efficacy of the bowel preparation | 1 hour after the colonoscopy
  Rating of the Boston Bowel Preparation Scale (BBPS) by the endoscopist

SECONDARY OUTCOMES:
Cecal intubation | 1 hour after the colonoscopy
  Ratio of successful cecal intubations in each study arm
Polyp and adenoma detection | 1 hour after the colonoscopy
  Ratio of polyps and adenomas detected in each study arm
Symptomatic hypoglycemia | 6 hours after finishing bowel preparation
  Each participant will report his/her experience in a questionnaire
Abdominal pain, nausea, hunger and bloating | 6 hours after finishing bowel preparation
  Each participant will rate his/her experience in an analogue visual scale
Adverse events | 30 days after the colonoscopy
  Description of all spontaneously reported adverse events.
Adherence to the planned bowel cleansing method (questionnaire) | 6 hours after finishing bowel preparation
  Each participant will rate his/her experience in a questionnaire.
Acceptability of the preparation (interference with work, leisure activities or sleep | 6 hours after finishing bowel preparation
  Each participant will rate his/her experience in a questionnaire.
Predictors of inadequate bowel preparation | Baseline
  Independent predictors will be identified by multivariate analysis

CONTACTS AND LOCATIONS:
Overall Officials: Marco Antonio Alvarez González, MD, PhD, Principal Investigator — Parc de Salut Mar
Locations (2):
- Spain (2):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital del Mar, Barcelona, Barcelona

REFERENCES:
- [Background] Taylor C, Schubert ML. Decreased efficacy of polyethylene glycol lavage solution (golytely) in the preparation of diabetic patients for outpatient colonoscopy: a prospective and blinded study. Am J Gastroenterol. 2001 Mar;96(3):710-4. doi: 10.1111/j.1572-0241.2001.03610.x. PMID 11280539
- [Background] Ozturk NA, Gokturk HS, Demir M, Erdogan D, Unler GK, Gur G, Yilmaz U. The effect of autonomous neuropathy on bowel preparation in type 2 diabetes mellitus. Int J Colorectal Dis. 2009 Dec;24(12):1407-12. doi: 10.1007/s00384-009-0757-4. Epub 2009 Jul 7. PMID 19582466
- [Background] Chung YW, Han DS, Park KH, Kim KO, Park CH, Hahn T, Yoo KS, Park SH, Kim JH, Park CK. Patient factors predictive of inadequate bowel preparation using polyethylene glycol: a prospective study in Korea. J Clin Gastroenterol. 2009 May-Jun;43(5):448-52. doi: 10.1097/MCG.0b013e3181662442. PMID 18978506
- [Derived] Alvarez-Gonzalez MA, Flores-Le Roux JA, Seoane A, Pedro-Botet J, Carot L, Fernandez-Clotet A, Raga A, Pantaleon MA, Barranco L, Bory F, Lorenzo-Zuniga V. Efficacy of a multifactorial strategy for bowel preparation in diabetic patients undergoing colonoscopy: a randomized trial. Endoscopy. 2016 Nov;48(11):1003-1009. doi: 10.1055/s-0042-111320. Epub 2016 Aug 4. PMID 27490086